CLINICAL TRIAL: NCT01099436
Title: A Phase III Randomized Trial With NEOadjuvant Chemotherapy (TAC) With or Without ZOledronic Acid for Patients With HER2- Negative Large Resectable or Locally Advanced Breast Cancer(NEO-ZOTAC)
Brief Title: Neo-Adjuvant Chemotherapy (TAC) With or Without Zoledronic Acid in Treating HER2-negative Breast Cancer Patients
Acronym: NEO-ZOTAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Borstkanker Onderzoek Groep (Network)
Collaborators: Dutch Cancer Society (Other); Amgen (Industry); Sanofi (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG-2010-01; CDR0000669246 (Registry Identifier: PDQ (Physician Data Query)); BOOG-NEO-ZOTAC (Other: BOOG); 2009-016932-11 (EudraCT Number)
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: HER2-negative breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Zoledronic Acid; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAC + Zoledronic acid (Experimental): six cycles of docetaxel (Taxotere®), Adriamycin® (endoxan) and Cyclofosfamide (TAC) and zoledronic acid (Zometa)
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Drug: zoledronic acid; Procedure: neoadjuvant therapy
- TAC (Active Comparator): six cycles of docetaxel (Taxotere®), Adriamycin® (endoxan) and Cyclofosfamide (TAC)
  Interventions: Drug: cyclophosphamide; Drug: docetaxel; Drug: doxorubicin hydrochloride; Procedure: neoadjuvant therapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: zoledronic acid
  Arms: TAC + Zoledronic acid
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, docetaxel, and zoledronic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether combination chemotherapy is more effective when given together with zoledronic acid in treating patients with breast cancer.

PURPOSE: This randomized phase III trial is studying giving doxorubicin hydrochloride together with cyclophosphamide and docetaxel to see how well it works with or without zoledronic acid in treating patients with large resectable or locally advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the value of neoadjuvant chemotherapy comprising doxorubicin hydrochloride, cyclophosphamide, and docetaxel with or without zoledronic acid in patients with HER2-negative large resectable or locally advanced breast cancer.

Secondary

* To correlate clinical response with pathological responses in both treatment arms.
* To evaluate the disease-free survival and overall survival of patients treated with this regimen.
* To evaluate the safety and tolerability of adding zoledronic acid to neoadjuvant chemotherapy.
* To evaluate heterogeneity of the ER/PR and HER2 measurement in core biopsy and the surgical specimen.

OUTLINE: Patients are randomized between 2 treatment arms.

* Arm I: Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV, and docetaxel IV on day 1. Patients also receive zoledronic acid IV over 15 minutes on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive doxorubicin hydrochloride IV, cyclophosphamide IV, and docetaxel IV as in arm I. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Large resectable or locally advanced disease

    * T2 (≥ 2 cm and positive lymph nodes), T2 (≥ 3 cm), ≥ T3, T4, any N, M0 disease
* Measurable disease (breast and/or lymph nodes)
* HER2-negative disease by core biopsy
* No evidence of distant metastases (M1)
* No prior breast cancer

PATIENT CHARACTERISTICS:

* Female
* Menopausal status unspecified
* WHO performance status 0-2
* Not pregnant or nursing
* WBC ≥ 3.0 x 10^9/L
* Neutrophil count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Bilirubin ≤ 1.5 times upper limit of normal (UNL)
* ALT and/or AST ≤ 2.5 times UNL
* Alkaline phosphatase ≤ 5 times UNL
* Creatinine clearance ≥ 50 mL/min
* Accessible for treatment and follow-up
* No previous malignancy within the past 5 years except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* No peripheral neuropathy > grade 2 (of any cause)
* No other serious diseases including recent myocardial infarction, clinical signs of cardiac failure, or clinically significant arrhythmias
* No poor dental health
* No known hypersensitivity reaction to any of the components of the treatment
* No medical or psychological condition that, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent

PRIOR CONCURRENT THERAPY:

* No prior breast surgery except for biopsy
* No prior chemotherapy or radiotherapy
* No prior bisphosphonates

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response after neoadjuvant chemotherapy with or without zoledronic | after surgery

SECONDARY OUTCOMES:
Correlation of clinical response with pathological responses of both treatment arms | after surgery
Disease-free survival | 3 and 5 years
Overall survival | 3 and 5 years
Safety and tolerability | during treatment
Heterogeneity of the ER/PR and HER2 measurement in core biopsy and the surgical specimen | at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Judith Kroep, MD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] de Groot S, Pijl H, Charehbili A, van de Ven S, Smit VTHBM, Meershoek-Klein Kranenbarg E, Heijns JB, van Warmerdam LJC, Kessels LW, Dercksen MW, Pepels MJAE, van Laarhoven HWM, Vriens BEPJ, Putter H, Fiocco M, Liefers GJ, van der Hoeven JJM, Nortier JWR, Kroep JR; Dutch Breast Cancer Research Group. Addition of zoledronic acid to neoadjuvant chemotherapy is not beneficial in patients with HER2-negative stage II/III breast cancer: 5-year survival analysis of the NEOZOTAC trial (BOOG 2010-01). Breast Cancer Res. 2019 Aug 28;21(1):97. doi: 10.1186/s13058-019-1180-6. PMID 31455425
- [Derived] de Groot S, Charehbili A, van Laarhoven HW, Mooyaart AL, Dekker-Ensink NG, van de Ven S, Janssen LG, Swen JJ, Smit VT, Heijns JB, Kessels LW, van der Straaten T, Bohringer S, Gelderblom H, van der Hoeven JJ, Guchelaar HJ, Pijl H, Kroep JR; Dutch Breast Cancer Research Group. Insulin-like growth factor 1 receptor expression and IGF1R 3129G > T polymorphism are associated with response to neoadjuvant chemotherapy in breast cancer patients: results from the NEOZOTAC trial (BOOG 2010-01). Breast Cancer Res. 2016 Jan 6;18(1):3. doi: 10.1186/s13058-015-0663-3. PMID 26738606
- See also: Clinical trial summary BOOG website — https://www.boogstudycenter.nl/studie/247/neo-zotac.html